CLINICAL TRIAL: NCT01652833
Title: Survey of Oncologists in Europe to Evaluate Their Knowledge of KRAS Testing
Brief Title: European Physician Survey of EGFR Inhibitor Prescribing Patterns
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20101121
Record Dates: First submitted 2012-06-05; First posted 2012-07-30 (Estimated); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Round 1: survey of 150 oncologists
  Interventions: Other: Physician Survey
- Round 2: survey of 150 oncologists approximately 12 months after round 1
  Interventions: Other: Physician Survey
- Round 3: survey of 150 oncologists approximately 24 months after round 1
  Interventions: Other: Physician Survey

INTERVENTIONS:
Other: Physician Survey — Eligible physicians will be contacted via telephone to perform the physician survey. A standardised questionnaire will be used to collect information about the physician's awareness of the correct indication and appropriate administration of Vectibix and the physician's experience in the administration of Vectibix treatment in the previous 6 months

SUMMARY:
To ensure the appropriate administration of Vectibix for the treatment of mCRC with wild-type KRAS in real-world practice, it is important to understand the awareness of practicing oncologists regarding the correct indication and appropriate administration of Vectibix. It is also critical to monitor changes in oncologists' awareness and practice between the different rounds of the study.

DETAILED DESCRIPTION:
The survey will be conducted for 3 rounds in months 0, 12, and 24 after the first interview.

Before the beginning of each round, a sampling list will be created by Amgen.

In each round of the survey, potential participating oncologists will be sampled from each country's sampling list through random sampling and reached through telephone, letter or email. During the initial contact, the oncologists will be assessed for their eligibility to participate in the study by using a standardized screening questionnaire.

The initial contact and screening of potential participating oncologists will continue until a total of 150 eligible oncologists agree to participate in each round. The number of oncologists sampled in each country will be proportional to the use of Vectibix in each country and the number of oncology physicians estimated to prescribe Vectibix. Each eligible oncologist can only participate in 1 of the 3 rounds of survey.

Study staff will then conduct the survey with each of the identified eligible oncologists over the telephone, using a standardized questionnaire. Information about their awareness of the correct indication and appropriate administration of Vectibix and their experience in the administration of Vectibix treatment in the previous 6 months will be collected. We will make every attempt to collect the correct information from participating oncologists. This may require at least two phone calls to allow an oncologist to review their notes in order to report the correct data.

ELIGIBILITY:
Physician Inclusion Criteria:

* Must be a practicing oncology specialist
* Must treat at least 3 new or continuing patients with metastatic colorectal cancer in the last quarter
* Must have prescribed Vectibix within the last 6 months to metastatic colorectal cancer patients

Exclusion Criteria:

* Must not have taken part in this study previously
* Must not have participated in Amgen study number 20101120.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physician's satisfying all of the eligibility criteria are eligible to be enrolled in the survey
Sampling Method: Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Proportion of oncologists who are aware of the correct indication of Vectibix, with regard to tumor KRAS status and who conduct a KRAS test prior to initiation of Vectibix treatment | Trend survey of physicians performed over 3 years
Proportion of oncologists who conduct a KRAS test prior to the initiation of Vectibix treatment | Trend survey of physicians performed over 3 years
Proportion of oncologists who administer Vectibix in mCRC patients with mutant KRAS tumors or with KRAS status unknown | Trend survey of physicians performed over 3 years
Proportion of oncologists who administer Vectibix simultaneously with oxaliplatin-containing chemotherapy in mCRC patients with mutant KRAS tumors or patients with tumor KRAS status unknown | Trend survey of physicians performed over 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com